CLINICAL TRIAL: NCT00599664
Title: Double-Blind, Placebo-Controlled, Two-Center, Pharmacokinetic Study Evaluating the Systemic Absorption and Safety of OMS201 in Subjects Undergoing Ureteroscopic Treatment of Unilateral Ureteral- or Renal Collecting System-Located Stones
Brief Title: Pharmacokinetic and Safety Study of OMS201 in Subjects Undergoing Ureteroscopic Treatment for Removal of Urinary Tract-Located Stones
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Omeros Corporation (Industry)
Responsible Party: Gregory Demopulos, MD, CMO, CEO, Omeros Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C07-001
Record Dates: First submitted 2007-12-26; First posted 2008-01-24 (Estimated); Last update posted 2010-04-30 (Estimated); Status verified 2010-04

CONDITIONS: Urinary Calculi; Urinary Stones; Urinary Tract Stones
Keywords: Urinary Calculi; Urinary Stones; Urinary Tract Stones; Calculi
MeSH Terms: conditions — Urinary Calculi; Calculi

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Drug
  Interventions: Drug: OMS201
- 2 (Placebo Comparator): Vehicle
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: OMS201 — OMS201 irrigation solution during surgery
  Arms: 1
Drug: Vehicle — Vehicle irrigation solution during surgery
  Arms: 2

SUMMARY:
Evaluate the safety and systemic absorption of OMS201 following exposure during ureteroscopy.

DETAILED DESCRIPTION:
OMS201 is being developed to facilitate endoscopy of the ureters and to reduce postoperative discomfort, such as pain, frequency, urgency and/or difficult urination following endoscopic surgery to remove a urinary tract stone.

ELIGIBILITY:
Inclusion Criteria:

* Subject is undergoing unilateral ureteroscopic removal of renal collecting system or ureteral stones located in the ureter with a maximum stone diameter of 12 mm, for which general anesthesia will be used.
* Subject's physical examination is within normal limits or examination is clinically non-significant for purposes of the study as determined by the Investigator, and subject is in good general health.
* Subject's laboratory evaluations are within normal limits or evaluations are clinically non-significant as determined by the Investigator.
* Female subject of childbearing potential who is using an effective method of birth control within at least 14 days prior to surgery and has a negative pregnancy test.
* Subject is at minimal risk from anesthesia and is classified according to the American Society of Anesthesiologists Physical Status Classification as either PS-1 or PS-2.
* Subject's body mass index is between 19 and 35, inclusive, based on the Body Mass Index Table.

Exclusion Criteria:

* Subject taking a prohibited medication.
* Subject who has had a renal transplant, has a single kidney or has evidence of a compromised renal function as measured by abnormal serum creatinine, as judged by the Investigator, or who has evidence of urinary tract infection, or has prior history of open or laparoscopic surgery, or any history of an ureteral stricture.
* Subject who has congenital anomalies that would engender an increased procedural safety risk such as ureteropelvic junction obstruction resulting in severely dilated renal pelvis, duplicated urinary collecting system, horseshoe kidney or vascular anomalies such as renal arteriovenous fistulas or papillary necrosis.
* Subject has bilateral renal or ureteral stones requiring concurrent ureteroscopic removal.
* Subject with clinically significant hypotension at Screening.
* Subject who has a present condition or history of any clinically significant uncontrolled gastrointestinal, cardiovascular, hepatic, renal, hematological, endocrine, neurological, psychiatric, connective tissue, respiratory or other medical disorder as determined by the Investigator.
* Subject on chronic diuretic use.
* Subject who has taken or used an investigational drug or device within 30 days prior to the day of surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-12; Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic | Day of Surgery

SECONDARY OUTCOMES:
Safety | Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Scott Houston, Study Director — Omeros Corporation
Locations (2):
- United States (2):
  - UC Irvine Medical Center, Orange, California
  - University of Texas Southwestern, Dallas, Texas